CLINICAL TRIAL: NCT05468099
Title: Mitigating Effect of Bioaerosols During Orthodontic Procedures: a Randomized Controlled Trial
Brief Title: Aerosol Generation in Dental Clinics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Pro00103510
Record Dates: First submitted 2022-07-19; First posted 2022-07-21 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Risk Reduction; Occupational Exposure; Dentist-Patient Transmission
Keywords: aerosol; bioaerosol; dentistry; orthodontics; saliva; nose
MeSH Terms: conditions — Risk Reduction Behavior | interventions — Povidone-Iodine

STUDY DESIGN:
Masking Description: Each participant and operator know the model which was assigned to them. The research assistant conducting the analysis is not able to identify the samples until analysis time.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Orthodontic debonding (Experimental)
  Interventions: Other: Chlorhexidine mouthwash and Povidone-Iodine; Device: High volume evacuator; Device: High volume evactuator and saliva ejector; Device: Local Exhaust System

INTERVENTIONS:
Other: Chlorhexidine mouthwash and Povidone-Iodine — Chlorhexidine mouth rinse which participants use for 20 seconds before procedure. Moreover, Povidone-Iodine nasal swabs are used to disinfect nostrils
Device: High volume evacuator — High volume evacuator held by assistant to capture dental spray
Device: High volume evactuator and saliva ejector — High volume evacuator and saliva ejector held by assistant to capture dental spray
Device: Local Exhaust System — Local exhaust system hovers above patient head to capture dental spray

SUMMARY:
The study examines 4 different methods to reduce dental bioaerosol spread in orthodontic procedures.

DETAILED DESCRIPTION:
We aim to examine 4 different methods to reduce dental aerosol spread during orthodontic procedures. These methods are: 1) high-volume evacuator, 2) high-volume evacuator and saliva ejector 3) Local Exhaust System 4) disinfection with povidone-iodine nasal swabs and chlorhexidine mouthwash.

ELIGIBILITY:
Inclusion Criteria:

* Orthodontic debonding being performed
* Acceptance to participate in the study and provide required saliva and nasal samples

Exclusion Criteria:

* Refusal to participate
* Refusal to provide saliva/nasal swab samples
* Allergy to Chlorhexidine gluconate
* Allergy to Povidone-Iodine

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2022-03-29 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Particle concentration measurements across the 4 different types of interventions | During procedure
Mass concentration measurements across the 4 different types of interventions | During procedure
Bioaerosol measurement from the tracked sources | During procedure
  Sources include patient, operator and assistant saliva and nasal secretions, preprocedural ambient air, dental unit waterline

SECONDARY OUTCOMES:
Bacterial contamination on the inside surface of the mask of operators and assistants | During procedure
  Sources include patient, operator and assistant saliva and nasal secretions, preprocedural ambient air, dental unit waterline

CONTACTS AND LOCATIONS:
Overall Officials: Khaled Altabtbaei, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Yes
Bacteria rDNA sequences will be deposited in a public repository such as NCBI. Study protocol will be published along with the manuscript
Supporting Information: Study Protocol
Time Frame: Will be published as soon as